CLINICAL TRIAL: NCT01283880
Title: Renal Tubular Acidosis in Incident Renal Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: ML6919
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2011-01

CONDITIONS: Renal Transplant Disorder
Keywords: kidney; transplantation; metabolic acidosis; renal tubular acidosis; nephrocalcinosis
MeSH Terms: conditions — Acidosis; Acidosis, Renal Tubular; Nephrocalcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Metabolic acidosis is a common complication in incident renal transplant recipients. Protracted acidosis may be associated with osteoporosis, inflammation, negative protein balance and malnutrition, and last but not least may cause renal dysfunction. Preliminary data indicate an increased prevalence of nephrocalcinosis in renal transplant biopsies of incident patients presenting with metabolic acidosis. The present study aims (1)evaluate the prevalence and type of renal tubular acidosis (RTA) in incident renal transplant recipients and to identify clinical correlates and (2) to find associations between RTA, nephrolithiasis and nephrocalcinosis

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a single kidney transplant included in the protocol biopsy program.
* eGFR > 30 ml/min
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Evenepoel, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium